CLINICAL TRIAL: NCT00845715
Title: The Effect of Early Range of Motion on Clinical Outcomes, Patient Satisfaction, and Cuff Integrity Following Arthroscopic Rotator Cuff Repair. A Prospective Randomized Study.
Brief Title: Early Range of Motion Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Augustus Mazzocca, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-311-3; DF08-13
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Rotator Cuff Disease
Keywords: rotator cuff; rehabilitation; range of motion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early motion (Other)
  Interventions: Other: Early motion
- Standard motion (Other)
  Interventions: Other: Standard motion

INTERVENTIONS:
Other: Early motion — Early referral to physical therapy for range of motion (2 days post)
  Arms: Early motion
Other: Standard motion — Standard referral to physical therapy for range of motion (4 weeks post)
  Arms: Standard motion

SUMMARY:
The purpose of this study is to investigate whether there is a difference in the quality of life, ability to return to functioning (back to everyday life), the amount of experienced pain in patients who immediately move their shoulder versus patient who delay moving their shoulder after arthroscopic rotator cuff repair. We are also interested in whether there is a difference in the healing rates between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who are between 18 years and 70 years of age
* full thickness rotator cuff tear on ultrasound and MRI
* failed conservative management

Exclusion Criteria:

* concomitant pathology including massive rotator cuff tears that extend into the subscapularis or the teres minor and all co-existing labral pathology
* history of neuromuscular or degenerative disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | 6 month post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Augustus D Mazzocca, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States